CLINICAL TRIAL: NCT05692180
Title: Efficacy and Safety of Benralizumab in Paediatric Patients With Severe Eosinophilic Asthma (DOMINICA)
Brief Title: A Multicentre, Randomised, Double-blind, Parallel Group, Placebo-controlled, Time-to-first Asthma Exacerbation Phase III Efficacy and Safety Study of Benralizumab in Paediatric Patients With Severe Eosinophilic Asthma (DOMINICA)
Acronym: DOMINICA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3250C00024
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Asthma
Keywords: Eosinophilic asthma; Pediatric Patients; Severe asthma
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab (Experimental): Patients will receive Benralizumab as an active solution via a subcutaneous (SC) injection.
  Interventions: Drug: Benralizumab
- Placebo (Placebo Comparator): Patients will receive a matching solution of the placebo via SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benralizumab — Benralizumab active solution will be administered SC to the patients.
  Arms: Benralizumab
Drug: Placebo — Placebo solution will be administered SC to the patients.
  Arms: Placebo

SUMMARY:
A study to evaluate the efficacy and safety of benralizumab administered subcutaneously in patients ≥ 6 to < 18 years of age with severe eosinophilic asthma, including a well-documented history of asthma exacerbations and uncontrolled asthma receiving high-dose inhaled corticosteroid (ICS) plus at least one additional controller medication.

DETAILED DESCRIPTION:
A randomised, double-blind, parallel-group, placebo-controlled, time-to-first-asthma-exacerbation event study designed.

There will be a screening period of 2 months to allow adequate time for the eligibility criteria to be evaluated. The screening period may be reduced to not lesser than 4 weeks from Visit 2a. Furthermore, the Screening Period may be extended up to 12 weeks (or longer, if deemed necessary by the investigator), to accommodate treatment.

Visit 2 will be split into Part A (Visit 2a) and Part B (Visit 2b) to reassess eligibility prior to randomisation and first dose of study treatment administration.

Patients will be randomised 1:1 to receive benralizumab or placebo.

The treatment period will consist of 2 parts: double-blind (DB) treatment period and open-label extension (OLE) period.

The initial placebo-controlled, DB treatment period will be of variable duration. The minimum duration of treatment in the DB treatment period for each patient will be 16 weeks. Patient will continue in the DB treatment period until the patient experiences an exacerbation or the required number of events have been observed in the study, whichever occurs sooner.

All patients who experience an asthma exacerbation in the DB treatment period will be offered the opportunity to continue into the OLE period. The OLE period is intended to allow each patient at least 48 weeks in the ≥ 12 to < 18-year-old age group and at least 2 years (104 weeks) in the ≥6 to < 12-year-old age group of treatment with benralizumab.

An end-of-the-treatment visit will occur 8 weeks after the last dose in the OLE

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving assent (signing the assent form) to participate in the study. The caregiver of the patient must be capable of giving written informed consent for the patient's participation in the study. Consent and assent forms must be completed prior to any study-specific procedures.
* Patient and the caregiver (where applicable) must be willing to and be able to answer questionnaires that are part of the study procedures.
* Male or female patients aged ≥ 6 to < 18 years old.
* Patients with physician-diagnosed severe eosinophilic asthma for at least 12 months prior to Visit 1.
* Patients with a diagnosis of severe asthma confirmed, evaluated, and managed by the clinical site/site network for ≥ 6 months prior to Visit 1.
* Patients with an exacerbation history of asthma exacerbations (defined as a requirement for systemic corticosteroids and/or hospitalisation) within 12 months prior to Visit 1, OR,

  1. 2 asthma exacerbations (defined as a requirement for systemic corticosteroids and/or hospitalisation) per year within the 2 years prior to Visit 1 AND, one or more of the following:
  2. Currently on stable maintenance oral corticosteroids (OCS) used for at least 3 months prior to Visit 1, OR,
  3. At least one of the 2 exacerbations that occurred in the year prior to Visit 1 resulted in hospitalisation.
* Patients on well-documented, stable treatment for asthma with high dose ICS and at least one additional controller medication, such as long-acting β2 agonists (LABA), leukotriene receptor antagonists (LTRA), long-acting muscarinic antagonists (LAMA), or theophylline, since at least 6 months prior to Visit 1.
* Eosinophilic airway inflammation that is related to asthma characterised as eosinophilic in nature as indicated by peripheral blood eosinophil count of ≥ 300 cells/μL during screening OR a blood eosinophil count of 150 to 299 cells/μL and documentation of elevated eosinophils in bronchoalveolar lavage (BAL), sputum, or bronchial biopsy within the 2 years prior to Visit 1.
* ≥ 70% compliance with maintenance asthma medication during the screening period based on the Paediatric Asthma Symptom - Observer reported (PASO) or Asthma Daily Diary.
* At least 70% daily PASO or Asthma Daily Diary completion during the entire screening period, with at least 50% PASO or Asthma Daily Diary completion in the 14-day period prior to randomisation.
* Pre-BD FEV1 ≤ 95% of the predicted normal value or pre-BD FEV1/FVC ratio < 0.85 required at Visit 1. Patients with ≥ 25 % increase in pre-BD FEV1 value during the screening period will be screen failed.
* ACQ-IA ≥ 1.5 with no meaningful improvement (ACQ-IA change ≤ -0.5) between screening and Visit 2a.
* Body weight ≥ 15 kg.
* Females of childbearing potential (FOCBP) who are sexually active, as judged by the investigator, must commit to consistent and correct use of a highly effective method of contraception.

Exclusion Criteria:

* Clinically important pulmonary disease other than asthma or patients who have ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts.
* Life-threatening asthma.
* Asthma exacerbation requiring use of systemic corticosteroids or increase in maintenance dose of OCS within 2 weeks prior to Visit 2a or acute upper/lower respiratory infection that requires antibiotics or antiviral medication within 2 weeks prior to the first dose of the IP (Visit 2b).
* Any disorder that is not stable in the opinion of the investigator and could affect the safety of the patient during the study, influence the findings of the studies or their interpretations or impede the patient's ability to complete the entire duration of the study.
* History of anaphylaxis to any biologic therapy.
* Current malignancy, or history of malignancy.
* A helminth parasitic infection.
* Use of immunosuppressive medication.
* Receipt of immunoglobulin or blood products within 30 days prior to Visit 1.
* Receipt of any marketed or investigational biologic within 5 half-lives prior to Visit 1.
* Previously received benralizumab (MEDI-563).
* Participation in another interventional clinical study.
* Patients with known hypersensitivity to benralizumab or any of the excipients of the product.
* Currently pregnant, breastfeeding, or lactating females.
* Previous randomisation in the present study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2030-05-05 (Estimated); Study Completion 2032-05-16 (Estimated)

PRIMARY OUTCOMES:
Time to first asthma exacerbation | From Baseline (Week 0) to End of Treatment (EOT) in DB treatment period
  The effect of benralizumab on asthma exacerbations in paediatric and adolescent patients with uncontrolled asthma will be evaluated.

SECONDARY OUTCOMES:
Change from baseline, during the DB treatment period in Interviewer-Administered Version of the Asthma Control Questionnaire (ACQ-IA) | From Baseline (Week 0) to EOT in DB treatment period
  The effect of benralizumab on asthma control and symptoms will be assessed.
Change from baseline, during the DB treatment period in Asthma symptom score | From Baseline (Week 0) to EOT in DB treatment period
  The effect of benralizumab on asthma control and symptoms will be assessed.
Change from baseline, during the DB treatment period in rescue medication use | From Baseline (Week 0) to EOT in DB treatment period
  The effect of benralizumab on asthma control and symptoms will be assessed.
Change from baseline, during the DB treatment period in night-time awakenings due to asthma | From Baseline (Week 0) to EOT in DB treatment period
  The effect of benralizumab on asthma control and symptoms will be assessed.
Change from baseline, during the DB treatment period in peak expiratory flow (PEF) | From Baseline (Week 0) to EOT in DB treatment period
  The effect of benralizumab on asthma control and symptoms will be assessed.
Serum benralizumab trough concentration | During Day -7, Day 56, Day 112, every 16 weeks and at EOT DB treatment period
  The pharmacokinetics of benralizumab will be characterised.
Anti-benralizumab antibodies | During Day -7, Day 56, Day 112, every 16 weeks and at EOT DB treatment period
  The immunogenicity of benralizumab will be characterised.
Change from baseline, during the DB treatment period in Paediatric Asthma Quality of Life Questionnaire-Interviewer Administered (PAQLQ-IA) total score | From Baseline (Week 0) to EOT in DB treatment period
  The effect of benralizumab on asthma health-related quality of life will be assessed.
Change from baseline, during the DB treatment period, in spirometry, for pre-dose/pre-bronchodilator forced expiratory volume in one second (FEV1) | From Baseline (Week 0) to EOT in DB treatment period
  The effect of benralizumab on pulmonary function (FEV1) will be assessed.
Change from baseline, during the DB treatment period, in spirometry, for post-bronchodilator FEV1 | From Baseline (Week 0) to EOT in DB treatment period
  The effect of benralizumab on pulmonary function (FEV1) will be assessed.
The Annualised asthma exacerbation rate (AAER) in the DB treatment period | From Screening until the EOT double blind treatment period
  The asthma exacerbations reported during the DB treatment period of the study will be described.

OTHER OUTCOMES:
Number of patients with Adverse events (AEs) and Serious adverse events (SAEs) | From Screening period until EOT DB treatment period
  The safety and tolerability of benralizumab will be evaluated.
The AAER in the OLE period | From Week 0 until the EOT OLE period
  The annualised rate of severe exacerbations in the OLE period will be assessed.

CONTACTS AND LOCATIONS:
Locations (82):
- United States (27):
  - Research Site, Mobile, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Madera, California
  - Research Site, Torrance, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Owensboro, Kentucky
  - Research Site, Lafayette, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Glenn Dale, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ridgeland, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Brick, New Jersey
  - Research Site, Northfield, New Jersey
  - Research Site, The Bronx, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Charleston, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Morgantown, West Virginia
- Argentina (9):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Ciudad de Buenos Aire
  - Research Site, Florida
  - Research Site, Lobos
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Rosario
  - Research Site, San Juan Bautista
  - Research Site, Santa Fe
- Canada (5):
  - Research Site, Edmonton, Alberta
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- France (7):
  - Research Site, Créteil
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Rouen
  - Research Site, Toulouse
- Germany (2):
  - Research Site, Essen
  - Research Site, Wesel
- Italy (6):
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Pavia
  - Research Site, Ponte San Pietro
  - Research Site, Roma
  - Research Site, Verona
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Rzeszów
  - Research Site, Skarżysko-Kamienna
  - Research Site, Tarnów
- South Korea (3):
  - Research Site, Cheongju-si
  - Research Site, Junggu
  - Research Site, Seoul
- Spain (8):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Benalmádena
  - Research Site, Cartagena
  - Research Site, Esplugues de Llobregat
  - Research Site, Madrid
  - Research Site, Mérida
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home